CLINICAL TRIAL: NCT00419029
Title: Motivational Interviewing to Engage OEF/OIF Veterans in Mental Health Treatment
Brief Title: Motivational Interviewing to Engage Operations Enduring Freedom and Iraqi Freedom (OEF/OIF) Veterans in Mental Health Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen Seal, Principle Investigator, San Francisco Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MH 06-004
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Combat Disorders; Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders
Keywords: combat; depression; PTSD; substance abuse
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Depression; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): brief telephone check-in (no motivational interviewing)
  Interventions: Behavioral: control
- telephone-administered motivational interviewing (Experimental): motivational interviewing sessions
  Interventions: Behavioral: telephone-administered motivational interviewing

INTERVENTIONS:
Behavioral: telephone-administered motivational interviewing — telephone motivational interviewing
  Arms: telephone-administered motivational interviewing
Behavioral: control — brief telephone check-in (no motivational interviewing)
  Arms: control

SUMMARY:
The goal of this randomized controlled trial is to evaluate the efficacy of telephone-administered motivational interviewing (TAMI) to enhance VA mental health treatment engagement among veterans of Operations Enduring Freedom (OEF) and Iraqi Freedom (OIF) who screen positive for mental health disorders on telephone assessment. The investigators will evaluate whether TAMI results in improved mental health treatment engagement, decreased mental health symptoms and increased quality of life among OEF/OIF veterans with mental health disorders. The long-term aim of this study is to conduct rapid assessment and intervention to prevent chronic mental illness and associated disability among our newest generation of veterans.

DETAILED DESCRIPTION:
Project Background/Rationale: Recent reports suggest that a substantial proportion of OEF/OIF veterans suffer from one or more co-occurring mental health disorders, particularly post-traumatic stress disorder (PTSD), depression, and substance use disorders. Many newly returning veterans fail to initiate or complete an adequate course of mental health treatment largely owing to barriers that include inherent features of the mental illness, practical and logistical concerns, and stigma. Untreated mental illness threatens to produce functional and occupational disability as occurred with Vietnam-era veterans. Motivational Interviewing (MI) is an evidence-based, client-centered, therapeutic technique shown to enhance mental health treatment engagement in high-risk populations by helping patients explore and resolve barriers to care.

Project Objectives: The aims of this proposal are: (1) to evaluate the efficacy of telephone-administered motivational interviewing (TAMI) compared to telephone-administered informational support sessions (Control) to enhance mental health treatment initiation and retention among OEF/OIF veterans who screen positive for one or more mental health disorders; (2) to compare change in mental health symptoms and quality of life among veterans assigned to TAMI versus Control, and (3) to describe barriers to mental health treatment engagement among OEF/OIF veterans and assess the putative mechanism by which TAMI increases mental health treatment engagement.

Project Methods: The study is a two-arm randomized controlled trial. We will conduct telephone-administered psychometric screening for PTSD, depression, high-risk alcohol and substance use among 1,000 OEF/OIF veterans residing in Northern California. In addition, we will collect baseline data on sociodemographic and military service-related characteristics, VA and non-VA mental health treatment experiences, barriers and motivation to initiate and/or follow-up with VA mental health appointments. Approximately 300 OEF/OIF veterans screening positive for one or more mental health disorders will receive a referral to mental health treatment in their area and will be randomly assigned to either an initial TAMI session followed by two booster TAMI sessions at 1 and 3 months versus three informational support sessions balanced for time and attention. We will measure outcomes at baseline, one, three, and six months. We will test the hypotheses that OEF/OIF veterans receiving TAMI as compared to the Control condition will be more motivated and hence more likely to overcome barriers to initiate and attend follow-up VA mental health treatment appointments and will have greater improvements in mental health symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of OEF/OIF with service in Iraq or Afghanistan, or areas surrounding these combat theaters
* Military service separation date after 9/30/01
* Has a zip code that corresponds to a Northern California address and no plans to relocate
* May be contacted by telephone
* Must screen positive for one or more of the following: PTSD, depression, high-risk alcohol and/or illicit substance use to enroll in the randomized controlled trial.

Exclusion criteria:

* Veterans who served post-9/11/01 but who did not serve in Operation Enduring Freedom or Operation Iraqi Freedom
* In VA or non-VA mental health treatment currently
* Residing more than 60 miles from San Francisco VA or a Community-based outpatient clinic associated with San Francisco VA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of TAMI, the primary outcome is the binary distinction between those who make an initial phone call to the OEF/OIF Combat Case Manager to arrange for a mental health treatment appointment versus those who do not (Aim 1). | measured 6 months post last follow-up appointment

SECONDARY OUTCOMES:
the binary distinction between attending an initial or re-engagement VA mental health treatment appointment versus not | 6 months post last follow-up appointment
the total number of VA mental health treatment sessions attended | 6 months p ost last follow-up appointment
the proportion of sessions attended per those scheduled during the 6-month follow-up period | 6 months post last follow-up
change in mental health symptom scores between the TAMI and Control groups | last follow-up appointment
change in quality of life score from baseline at 1, 3, and 6 months. | last follow-up appointment

CONTACTS AND LOCATIONS:
Overall Officials: Karen H Seal, MD, MPH, Principal Investigator — San Francisco VA Medical Center, University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States